CLINICAL TRIAL: NCT01671254
Title: A Double-blind, Placebo-controlled Trial of a Dietary Supplement Containing Citrus Bioflavonoids and Vitamin E at 2 Doses in Conjunction With Fish Oil Supplementation in Hyperlipidemic Subjects
Brief Title: Effect of Citrus Bioflavonoids/Vitamin E in Conjunction With Fish Oil Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetaProteomics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: POT2-FMR-CT
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- FishOil + placebo (Active Comparator): Subjects in this arm receive fish oil (EPA/DHA Extra Strength) and placebo capsule
  Interventions: Dietary Supplement: FishOil; Dietary Supplement: placebo
- FishOil + CBE75 (Experimental): Subjects in this arm receive fish oil (EPA/DHA Extra Strength) and citrus bioflavonoids+vitamin E (CBE)(75 mg/capsule/day)
  Interventions: Dietary Supplement: FishOil; Dietary Supplement: CBE75
- FishOil + CBE150 (Experimental): Subjects in this arm receive fish oil (EPA/DHA Extra Strength) and CBE (150 mg/capsule/day)
  Interventions: Dietary Supplement: FishOil; Dietary Supplement: CBE150

INTERVENTIONS:
Dietary Supplement: FishOil
Dietary Supplement: CBE75
  Arms: FishOil + CBE75
Dietary Supplement: CBE150
  Arms: FishOil + CBE150
Dietary Supplement: placebo
  Arms: FishOil + placebo

SUMMARY:
The purpose of this 8-week intervention trial is to investigate the effect of a dietary supplement (containing citrus bioflavonoids and vitamin E) plus fish oil supplementation in healthy hyperlipidemic subjects

ELIGIBILITY:
Inclusion Criteria:

* men and women ≥ 18 and ≤ 72 years old
* generally healthy
* BMI > 18 and < 38
* LDL cholesterol ≥ 130 mg/dl and < 270 mg/dl
* triglycerides ≥ 150 mg/dl and < 400 mg/dl
* ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* use of nutritional supplements and medical foods for dyslipidemia within 30 days prior to the study
* use of omega-3 fatty acid dietary supplements within 30 days prior to the study
* use of prescription HMG-CoA reductase inhibitors, bile acid sequestrants, fibrates, cholesterol absorption blocking agents, or niacin
* use of prescription medications and/or nonprescription medications for acute and semi-acute medical conditions
* history of cardiovascular disease, type i diabetes, autoimmune disease, liver or kidney disease, malignancy, and serious mental illness.
* known infection with HIB, TB, hepatitis B or hepatitis C
* history of allergy or intolerance to study products
* smoking, use of nicotine-containing products, or use of drugs of abuse 30 days prior to the study
* history of regular intake of > 14 alcoholic drinks per week for females and > 21 drinks per week for males

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | Baseline, 8 weeks
  Change in LDL cholesterol level at the end of 8 weeks

SECONDARY OUTCOMES:
Triglyceride | Baseline, 8 weeks
  Change in triglyceride level at the end of 8 weeks.
oxLDL | Baseline, 8 weeks
  Change in oxidized LDL level at the end of 8 weeks.
Total cholesterol | Baseline, 8 weeks
  Change in total cholesterol level at the end of 8 weeks.
HDL cholesterol | Baseline, 8 weeks
  Change in HDL cholesterol level at the end of 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Lamb, MD, Principal Investigator — MetaProteomics / Metagenics / FMRC
Locations (1):
- Functional Medicine Research Center, Gig Harbor, Washington, United States